CLINICAL TRIAL: NCT00466492
Title: Advantages and Disadvantages of Long Term Sedation in ICU Patients
Brief Title: Advantages and Disadvantages of Long Term Sedation in Intensive Care Unit Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Thomas Strøm, Anaesthesiologic-intensive unit, Odens University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-6-06
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2009-06

CONDITIONS: Critical Illness; Length of Stay; Respiration, Artificial; Intensive Care Units
Keywords: Drug Administration Schedule; Intensive Care Units; Length of Stay; Respiration, Artificial; Stress Disorders, Post-Traumatic/etiology/*psychology; Critical Illness/*psychology; Pneumonia/prevention & control; Hypnotics and Sedatives/*administration & dosage
MeSH Terms: conditions — Critical Illness; Respiratory Aspiration; Stress Disorders, Traumatic; Pneumonia | interventions — Wake protein, Drosophila; Critical Care; hemoglobin Denmark Hill; Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No sedatation intervention (Other): The intervention group is the normal care in our institution, the control group is the golden standard
  Interventions: Procedure: Sedation or no sedation during mechanical ventilation

INTERVENTIONS:
Procedure: Sedation or no sedation during mechanical ventilation — No sedation to critically ill patients
  Other Names: Awake; intensive care; Denmark; Mechanical ventilation

SUMMARY:
The purpose of the study is to determine whether sedation of the critical ill patient prolongs the time receiving mechanical ventilation.

DETAILED DESCRIPTION:
The golden standard is to sedate critical ill patients receiving mechanical ventilation with daily wake up trials. This is shown to reduce the time receiving mechanical ventilation compared to no wake up trials.

We would like to study whether no sedation but only analgesics administered as bolus doses, reduce the time receiving mechanical ventilation. The study is planned as a randomised prospective study, not blinded. The control group is patients receiving sedation with daily wake up trials. The intervention group is not sedated, but receives bolus doses of analgesics (morphine). The endpoint is the time spend receiving mechanical ventilation, lengths of stay on the intensive care unit, and total lengths of stay on the hospital.

We also examine the frequency of ventilator associated pneumonia and CT scans of cerebrum. Also we would like to examine the long term psychological effects of sedation, we plan to send some of the patients to a post traumatic stress screening. The effect on the next of kin we plan to study with a questionnaire. As a last thing we would like to study the workload on the nurses.

ELIGIBILITY:
Inclusion Criteria:

* Intubated receiving mechanical ventilation
* Expected to remain intubated more than 24 hours
* Over 18 years

Exclusion Criteria:

* Raised intracranial pressure
* Pregnant
* Treatment with muscle relaxants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Time receiving mechanical ventilation, total intensive care and hospital length of stay.

SECONDARY OUTCOMES:
The frequency of VAP, CTC. The amount of Post Traumatic Stress after 6 month. The patients families experience. The workload on the nurses | VAP and CTC during hospital stay. PTSD 1-2 years after the primary stay

CONTACTS AND LOCATIONS:
Overall Officials: Palle Toft, Professor, Study Chair — Institute of Clinical Research
Locations (1):
- Anaesthesiologic-intensive Care Department, Odense University Hospital, Odense C, Odense C, Denmark

REFERENCES:
- [Result] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184
- [Result] Kress JP, Gehlbach B, Lacy M, Pliskin N, Pohlman AS, Hall JB. The long-term psychological effects of daily sedative interruption on critically ill patients. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1457-61. doi: 10.1164/rccm.200303-455OC. Epub 2003 Oct 2. PMID 14525802
- [Result] Schweickert WD, Gehlbach BK, Pohlman AS, Hall JB, Kress JP. Daily interruption of sedative infusions and complications of critical illness in mechanically ventilated patients. Crit Care Med. 2004 Jun;32(6):1272-6. doi: 10.1097/01.ccm.0000127263.54807.79. PMID 15187505
- [Derived] Strom T, Stylsvig M, Toft P. Long-term psychological effects of a no-sedation protocol in critically ill patients. Crit Care. 2011;15(6):R293. doi: 10.1186/cc10586. Epub 2011 Dec 13. PMID 22166673
- [Derived] Strom T, Johansen RR, Prahl JO, Toft P. Sedation and renal impairment in critically ill patients: a post hoc analysis of a randomized trial. Crit Care. 2011;15(3):R119. doi: 10.1186/cc10218. Epub 2011 May 4. PMID 21542927
- [Derived] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- See also: Link to the published paper — http://www.thelancet.com/journals/lancet/article/PIIS0140-6736(09)62072-9/abstract